CLINICAL TRIAL: NCT00059553
Title: Activity-Dependent Plasticity After Spinal Cord Injury
Brief Title: Retraining Walking After Spinal Cord Injury
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K01HD001348 (NIH)
Record Dates: First submitted 2003-04-28; First posted 2003-04-29 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2005-08

CONDITIONS: Spinal Cord Injuries; Quadriplegia; Paraplegia; Central Cord Syndrome; Brown-Sequard Syndrome
Keywords: spinal cord injury; walking; training; treadmill; incomplete spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Paraplegia; Central Cord Syndrome; Brown-Sequard Syndrome

INTERVENTIONS:
Behavioral: Locomotor treadmill training with body weight support

SUMMARY:
Incomplete spinal cord injury often results in difficulty walking. Training on a treadmill with body weight support may improve walking ability after spinal cord injury. The purpose of this study is to examine the effect of treadmill speed on spinal cord function and walking performance.

DETAILED DESCRIPTION:
Conventional rehabilitation following spinal cord injury (SCI) emphasizes functional gains through strengthening and compensation, using braces and assistive devices to achieve mobility. Rehabilitation practice using compensatory approaches is based on the prevailing assumption that neural recovery is not possible following SCI.

Recent evidence contradicts this assumption. Stimulated by the proper activation of peripheral afferents associated with walking, neuronal circuits may reorganize by strengthening of existing and previously inactive descending connections and local neural circuits. New approaches to locomotor recovery after SCI utilize sensory information related to locomotion to improve treadmill and overground walking.

Locomotor training velocity may be a critical, task-specific, and activity-dependent parameter affording appropriate phasic, afferent input to the neural system and promoting neural plasticity. The purpose of this study is to evaluate the effects of training velocity in a long-term locomotor training program on both neurophysiological and behavioral plasticity in individuals with incomplete SCI.

Sixteen patients with incomplete SCI will be recruited to participate in this study. Baseline evaluations will include American Spinal Injury Association classification, rate-sensitive depression, phase-dependent H-reflex modulation at self-selected and fast overground walking velocities, and MRI of the spine. Patients will wear a step activity monitor for a 48-hour period, quantifying baseline walking activity level.

All patients will participate in a locomotor training program. Patients will be randomly assigned to either training at self-selected treadmill velocity or at a normal walking velocity. Patients will have 45 training sessions over 9 weeks. Each training session will include 30 minutes of walking. Interim testing of rated depression, spatial-temporal parameters of walking, MRI, and walking activity will occur through the 9-week training period. Post-testing will occur within 2 days of the last training session and at a 1 month after completion of the training. During the month following long-term training, patients will be instructed to return to their self-selected routine activities of daily living.

ELIGIBILITY:
Inclusion criteria:

* First time spinal cord injury (SCI) from trauma, vascular, or orthopedic pathology at cervical or thoracic levels
* Category C or D SCI as defined by the American Spinal Injury Association (ASIA) Impairment Scale
* 1 to 3 years post-SCI
* Ability to walk independently a minimum of 40 feet with or without an assistive device
* Currently spending a minimum of 30 minutes per day walking
* No change in anti-spasticity medication during the study
* Medically stable
* Participant's personal physician must verify the participant's medical status

Exclusion criteria:

* Bladder infection, decubiti, osteoporosis, cardiopulmonary disease, pain, or other significant medical complications that would prohibit or interfere with training and testing of walking function or alter compliance with a training protocol
* Currently participating in a rehabilitation program or another research protocol that could interfere or influence the outcome measures of the current study
* Congenital SCI (e.g., Chiari malformation, myelomeningocele, intraspinal neoplasm, Frederich's ataxia)
* Other degenerative spinal disorders (e.g., spinocerebellar degeneration, syringomyelia) that may complicate the treatment or evaluation procedures

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16
Dates: Start 2000-05; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Behrman, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Behrman AL, Harkema SJ. Locomotor training after human spinal cord injury: a series of case studies. Phys Ther. 2000 Jul;80(7):688-700. PMID 10869131
- [Background] Barbeau H, Norman K, Fung J, Visintin M, Ladouceur M. Does neurorehabilitation play a role in the recovery of walking in neurological populations? Ann N Y Acad Sci. 1998 Nov 16;860:377-92. doi: 10.1111/j.1749-6632.1998.tb09063.x. PMID 9928326
- See also: Departmental Website for Principal Investigator — http://pt.phhp.ufl.edu/behrman.html
- See also: Website for Principal Investigator in Rehabilitation Science PhD Program — http://pt.phhp.ufl.edu/rsd.html